CLINICAL TRIAL: NCT04093986
Title: Hydroxyurea Exposure Limiting Pregnancy and Follow-Up Lactation
Acronym: HELPFUL
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Connecticut (Other); University of Colorado, Denver (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Duke University (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: HELPFUL
Record Dates: First submitted 2019-08-22; First posted 2019-09-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective Chart Review: Medical record chart review of women seen previously for clinical care prior to June 20, 2019 at participating institutions with SCD and hydroxyurea exposure during gestation or lactation will be identified by healthcare providers.
  Interventions: Other: Chart Review
- Participant Survey and Retrospective Chart Review: Participants providing their medical records without the assistance of a health care provider will be asked to complete a questionnaire through REDCap and will have the option to upload their deidentified medical records if they are available.
  Interventions: Other: Chart Review; Other: Survey

INTERVENTIONS:
Other: Chart Review — Medical records or data available from previous clinical care prior to June 20, 2019 about pregnancy and breastfeeding outcomes, both for babies with hydroxyurea exposure and other babies by these same women.
Other: Survey — Women who choose to participate directly and provide information in survey format will receive a brief survey and the option to upload their medical records (if available) into Cincinnati Children's maintained REDCap database.
  Groups: Participant Survey and Retrospective Chart Review

SUMMARY:
The purpose of this research study is to document and understand the effects of hydroxyurea exposure for women with SCD and their babies, during both gestation and lactation.

DETAILED DESCRIPTION:
Hydroxyurea (hydroxycarbamide) is the primary disease-modifying therapy for individuals with sickle cell disease (SCD) and is both US FDA- and EMA-approved for SCD treatment. Decades of research have documented that hydroxyurea reduces morbidity and mortality for affected patients. Although its primary mechanism of action for SCD is the induction of fetal hemoglobin (HbF) that prevents erythrocyte sickling, hydroxyurea is also a ribonucleotide reductase inhibitor with dose-dependent cytotoxic effects. Based on laboratory data, hydroxyurea is considered to be a potential human mutagen, clastogen, teratogen, and even carcinogen. However, most of these are theoretical human risks; for example, teratogenic effects of hydroxyurea are based on in vitro cellular data and supra-pharmacological dosing of animals, with no documented abnormalities in humans. Despite the lack of in vivo human data, the package insert for hydroxyurea, sold as either Hydrea® or Droxia® (Bristol-Myers Squibb), or as Siklos® (Addmedica) lists both pregnancy and lactation as contraindications for treatment.

This contraindication label is critically important, since women with SCD frequently have high-risk pregnancies throughout gestation, with increased morbidity and mortality for both the mother and baby. Acute clinical complications for the mother occur commonly during gestation, while placental insufficiency through repeated infarctions also leads to increased fetal morbidity. Protection of the mother's health during pregnancy is therefore a high priority, which historically has been aided by judicious use of transfusions and management by a multidisciplinary healthcare team. In the current era, many women with SCD of child-bearing age are taking daily oral hydroxyurea with an excellent treatment effect, so its forced discontinuation around the time of pregnancy represents cessation of effective therapy. Abrupt withdrawal of hydroxyurea is typically deleterious and may not be justified in this setting. Numerous published case reports and small series have described the safe use of hydroxyurea as anti-neoplastic therapy during pregnancy in women with cancer; moreover, anecdotal experience of >100 pregnancies with hydroxyurea exposure did not document any teratogenicity.

Based on the importance of determining the actual risks and benefits of continuing hydroxyurea as disease-modifying therapy during pregnancy to protect both mothers and babies, and the lack of documented in vivo data, the safety of hydroxyurea during gestation and subsequent lactation was recently identified as an important knowledge gap by the NHLBI evidence-based SCD guidelines. Further data collection is needed regarding the actual effects of hydroxyurea for women with SCD during both pregnancy and while breastfeeding. Accordingly, we will conduct a multinational research project to retrospectively capture known human exposures to hydroxyurea in the setting of SCD, which have occurred during gestation and/or lactation, to elucidate the outcomes for the mothers and their babies. Those outcomes will be compared to pregnancies in these same women without hydroxyurea exposure.

ELIGIBILITY:
Inclusion Criteria:

* Medical records or data available from previous clinical care prior to June 20, 2019 of pregnant females with SCD, including women who miscarried, had a still birth, or completed labor at any gestational stage, with any hydroxyurea exposure during either pregnancy and/or while breastfeeding.
* Medical records or data available from previous clinical care prior to June 20, 2019 about pregnancy and breastfeeding outcomes, both for babies with hydroxyurea exposure and other babies by these same women.

Exclusion Criteria:

* Unavailable medical records or lack of information about hydroxyurea exposure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical and laboratory data on up to 200 women with SCD with hydroxyurea exposure during either gestation or lactation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
How long pregnant women with Sickle Cell Disease (SCD) were exposed to Hydroxyurea. | Through completion of pregnancy, an average of 2 years
  Obtain data on length of time women with SCD were exposed to Hydroxyurea prior to pregnancy, during pregnancy, and after pregnancy.
Dose of hydroxyurea taken during pregnancy. | Through completion of pregnancy, an average of 2 years
  Obtain data on the dose of Hydroxyurea taken prior to conception, during and after pregnancy.
How long infants were exposed to Hydroxyurea. | Through study completion, an average of 2 years
  Obtain data on length of time infants were exposed to Hydroxyurea during gestation and while breastfeeding.
Dose of hydroxyurea exposure in infants. | Through study completion, an average of 2 years
  Obtain data on the dose of Hydroxyurea taken by mother during gestation and while breastfeeding infant.
Health outcomes of infants exposed to Hydroxyurea. | Through study completion, an average of 2 years
  Obtain data on the health of infant after exposure to Hydroxyurea during gestation and while breastfeeding including any complications of mother's pregnancy or delivery as well as any congenital malformations or medical conditions in infancy.
Pregnancy in Sickle Cell Disease (SCD). | Start of pregnancy until June 2019
  Compare pregnancy and delivery complications in women with SCD exposed to Hydroxyurea to pregnancy and delivery complications in women with SCD without Hydroxyurea exposure.
Comparative analysis of congenital malformations or medical conditions in infants | Through study completion, an average of 2 years
  Compare the rate of congenital malformations and/or medical conditions in infants exposed to hydroxyurea during gestation and breastfeeding to the rate of these events in infants without hydroxyurea exposure, with data collected descriptively by self-report or chart review as applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States